CLINICAL TRIAL: NCT01785446
Title: Effect of Dexmedetomidine on Cisatracurium Infusion and Sufentanil Consumption and Its Variations in Different Age Groups, Using a Closed Loop Computer Controlled System.
Brief Title: Study of Cisatracurium and Sufentanil Consumption Using a Closed Loop Computer Control Infusion System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Shehzaad Joomye (Unknown); Haiyun Wang (Unknown); Donglai Yan (Unknown)
Responsible Party: Principal Investigator, Guolin Wang, MD, PhD, Professor, M.D. PhD. Professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Cis-123
Record Dates: First submitted 2013-02-04; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: The Intraoperative Effect of Dexmedetomidine on Cisatracurium Infusion Consumption and Its Recovery Index.; Effect of Dexmedetomidine on Sufentanil Consumption.; Quantitative Analysis of Cisatracurium Infusion Requirements, Sufentanil Consumption and Recovery Index in Different Age Groups.
Keywords: Dexmedetomidine; Cisatracurion infusion; Sufentanil; Recovery Index; Closed loop computer control system
MeSH Terms: interventions — Dexmedetomidine; cisatracurium; Sufentanil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- P 1 (Active Comparator): In this group patients were aged from 20 to 45. Propofol infusion was used to maintain Bispectral Index (BIS) between 45 and 55.
  Intermittent doses of sufentanil 10-20 microgram were given intra-operatively on a required basis.
  Interventions: Drug: Consumption of cisatracurium and sufentanil in different age groups.
- P 2 (Active Comparator): In this group patients were aged from 46 to 65. Propofol infusion was used to maintain Bispectral Index (BIS) between 45 and 55.
  Intermittent doses of sufentanil 10-20 microgram were given intra-operatively on a required basis.
  Interventions: Drug: Effect of dexmedetomidine on cisatracurium and sufentanil consumption; Drug: Consumption of cisatracurium and sufentanil in different age groups.
- P 3 (Active Comparator): In this group patients were aged from 66 to 85. Propofol infusion was used to maintain Bispectral Index (BIS) between 45 and 55.
  Intermittent doses of sufentanil 10-20 microgram were given intra-operatively on a required basis.
  Interventions: Drug: Consumption of cisatracurium and sufentanil in different age groups.
- D (Active Comparator): In this group patients were aged from 46to 65. Propofol infusion was used to maintain Bispectral Index (BIS) between 45 and 55.
  Dexmedetomidine infusion is started at induction,a bolus dose of 0.5 µg/kg is given over the first hour which is followed by infusion of 0.4 µg/kg/hr.
  Intermittent doses of sufentanil 10-20 microgram were given intra-operatively on a required basis.
  Interventions: Drug: Effect of dexmedetomidine on cisatracurium and sufentanil consumption

INTERVENTIONS:
Drug: Effect of dexmedetomidine on cisatracurium and sufentanil consumption — In this intervention we compared the cisatracurium consumption, recovery index and sufentanil consumption between P2 and D. The reason we are comparing patients in group D with P2 is that because they belong to the same age group.
  Other Names: Dexmedetomidine
  Arms: D; P 2
Drug: Consumption of cisatracurium and sufentanil in different age groups. — For this intervention, we compared the cisatracurium consumption, refractory index and sufentanil consumption between group P1, P2 and P3.
  Arms: P 1; P 2; P 3

SUMMARY:
The purpose of this study is to:

* determine the effect of dexmedetomidine on cisatracurium infusion requirements and sufentanil consumption.
* analyze the cisatracurium infusion requirements and sufentanil consumption in different age groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1 and 2.
* Consent approval written and oral.
* Patients scheduled for elective abdominal surgery under general anesthesia.

Exclusion Criteria:

* Patients with neuromuscular disorders.
* Patients with history of stroke, flaccid paralysis or other neurological disorders.
* Significant renal, hepatic or cardiac dysfunction.
* Consent refusal.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Cisatracurium infusion consumption. | At the time of surgery
  Measurements were done during the operation. Cisatracurium infusion was controlled a closed loop computer system. The degree of neuromuscular blockage was assessed every 20 seconds throughout the procedure using the train of four testing. It was done by counting the number and amplitude of twitches evoked after electrical stimulus and the rate of infusion maintained itself at the low rate of 0.20µg/kg/min as long as the T1 response is less than 1%. When the T1 > 1%, the rate of infusion would automatically increase to 5.0 µg/kg/min until T1 < 1%, after which the infusion rate would fall back to 0.20µg/kg/min. The controlled infusion described above administered small doses of cisatracurium intra-operatively to maintain a muscle relaxation of more than 99%. The system saved the time and amount of drug given throughout the operation, from which the consumption was calculated in µg/kg/min.

SECONDARY OUTCOMES:
Sufentanil consumption. | At the time of operation.
  Analgesia was maintained by intermittent bolus dose of 10-20 µg of Sufentanil when the pulse and blood pressure would increase by more than 20% of the baseline, and BIS in the required range, as this would indicate an increase perception of pain but adequate anaesthesia. Sufentanil consumption was calculated for each patient in µg/kg/hr and the length of the operation was determined as from induction to the time of skin closure.

OTHER OUTCOMES:
Recovery Index | 30 minutes post-operative.
  Recovery Index, time for the Train-Of-Four (TOF) value to increase from 25% to 75%, was measured in each patient who completed the study. Its measurements were recorded in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD, PhD, Professor, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Joomye S, Yan D, Wang H, Zhou G, Wang G. Consumption of Cisatracurium in different age groups, using a closed loop computer controlled system. BMC Anesthesiol. 2014 Apr 21;14:29. doi: 10.1186/1471-2253-14-29. eCollection 2014. PMID 24745306